CLINICAL TRIAL: NCT02124356
Title: Functional Performance Following Emergency High-risk Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Morten Tange Kristensen, Seniorresearcher, Hvidovre University Hospital
Other Study IDs: HH-AHA-FYS-01; H-2-2014-FSP31 (Registry Identifier: Regional Ethics Committee)
Record Dates: First submitted 2014-04-23; First posted 2014-04-28 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-10

CONDITIONS: Emergency High-risk Abdominal Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Emergency High-risk Abdominal Surgery
  Interventions: Other: Evaluation of functional performance

INTERVENTIONS:
Other: Evaluation of functional performance

SUMMARY:
Emergency abdominal surgery is associated with high mortality rates, multiple postoperative complications and prolonged duration of hospital admission. The purpose of this study is to examine the postoperative functional performance in patients undergoing Emergency High-risk Abdominal Surgery. The hypothesis is that the study can describe the patient population in relation to postoperative functioning, degree of inactivity and the factors that limit mobility.

ELIGIBILITY:
Inclusion Criteria:

* Patients (19 years and older) undergoing emergency laparotomy or laparoscopy (inclusive reoperations after elective surgery).

Exclusion Criteria:

* Patients undergoing minor emergency operations (uncomplicated appendectomy, laparoscopic cholecystectomy, diagnostic laparoscopy or laparotomy without intervention)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (19 years and older) undergoing Emergency High-risk Abdominal Surgery at the Hvidovre University Hospital.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Basic mobility evaluated by the Cumulated Ambulation Score (CAS) | Daily on postoperative day 1 to 7 and at discharge from the hospital (average length of stay is: 14 days).
  Factors that limit independency in basic mobility will be evaluated on a daily basis.

SECONDARY OUTCOMES:
Physical activity assessment with accelerometer (ActivePAL) | Daily on postoperative day 1 to 7.
Visual Analog Scale (VAS) | Daily on postoperative day 1 to 7 and at discharge from the hospital (average length of stay is: 14 days).
  VAS is a self-reported measure of pain intensity.
Assessment of Motor and Process Skills (AMPS) | One time at postoperative day 4.
  AMPS measures a person's performance capacity for activities of daily living (ADL) and/or independent living.

OTHER OUTCOMES:
New Mobility Score (NMS) | At inclusion/baseline
  NMS is a measure of pre-hospital functional level.

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark